CLINICAL TRIAL: NCT05641948
Title: Radiofrequency Denervation and Brain Structure, Function And Connectivity In Chronic Low Back Pain Patients
Brief Title: Radiofrequency Denervation and Brain Imaging
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-078-22
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain, Mechanical
Keywords: Neuroimaging; Radiofrequency denervation
MeSH Terms: conditions — Low Back Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Back Pain: In this prospective observational study, patients with chronic low back pain, scheduled for possible treatment with radiofrequency denervation (RFD), will be recruited from the NHS Grampian pain clinic. In the clinical pathway, patients will undergo a diagnostic medial branch nerve block (MBB). The outcome of this test determines if they are suitable for RFD. For this study, patients will be recruited from the clinics before the MBB. They will have both clinical assessments of pain levels and quality of life and a brain scan at three time intervals - baseline before the diagnostic nerve block, after diagnostic nerve block and 3 months after RFD. The final eligibility for the study is confirmed after the diagnostic block.
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — Participants will undergo brain MRI scan at 3 intervals

SUMMARY:
The goal of this observational study is to learn about changes in brain and its activity of following radiofrequency denervation treatment for chronic low back pain. The main question it aims to answer are:

* report the magnitude of the brain changes following radiofrequency treatment for low back pain.
* identify changes unique to radiofrequency treatment

Patients with nociceptive type low back pain of moderate to severe intensity will be identified to undergo radiofrequency treatment. They will have 3 MRI scans - Baseline, after the diagnostic injections and 3 months after radiofrequency treatment. They will also fill questions relating to their pain, disability and health related quality of life.

DETAILED DESCRIPTION:
Low back pain is one of the most common pain conditions and is the leading cause of years lived with disability. The management is challenging due to the heterogeneity of clinical presentation and includes self-management, pain killers, targeted injections as well as pain management programs. Brain MRI scans have identified networks of brain regions and changes in their activity in chronic low back pain (cLBP) patients. The scans have also been used to explore treatment-induced changes in brain and its activity. Radiofrequency denervation (RFD) of medial branch nerves is a NICE recommended treatment for a sub-group of cLBP sufferers. There are inter-individual variations in the response to RFD, which have been difficult to predict. The brain MRI scans can be used to better understand the effects of RFD on brain structure and function, and to predict those most likely to benefit from the interventions. So, we propose pilot study to investigate brain regions, their patterns and change after RFD treatment in this subgroup of cLBP sufferers. Eligible patients will have 3 brain MRI scans at various time intervals - Baseline, after nerve block and after RFD.

These brain scans will be analysed to provide the foundations for new studies such as improved selection of patients most likely to benefit from the treatment; improved understanding of mechanisms of the RFD treatment; and develop objective measurements that could be used in future trials of pain treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Chronic moderate to severe cLBP (defined by average pain intensity of ≥ 4 in the 11 point Numerical Pain rating scale and a minimum duration of 1 year)
* Identified by clinical team as suitable for RFD pathway
* Predominantly nociceptive pain (as defined by PainDetect score ≤12)
* Stable on current analgesic regime
* Able to communicate in English
* Has the capacity to and agrees to give informed consent for participation in the study
* Positive response to a single diagnostic MBB with 1 ml or less of local anaesthetic (bupivacaine 0.5%) at each level. (a positive response is defined as ≥80% pain relief at 3 hours, based on patient reported assessment)

Exclusion Criteria:

* Any patient whose physical condition will preclude them from lying still for the duration of the brain scan.
* Contraindication to magnetic resonance scanning such as an implantable cardiac device.
* Women who are, or may be, pregnant. (Pregnant patients do not undergo pain procedures under radiological guidance as per routine clinical care)
* Significant anxiety and depression (as defined by HADS score ≥ 9)
* Clinical suspicion that alternative diagnosis is the reason for LBP
* Presence of chronic primary pain conditions (Fibromyalgia, chronic widespread pain, Complex Regional Pain Syndrome, Chronic Primary Headache, Orofacial pain, Chronic primary visceral pian and Chronic Primary musculoskeletal pain as defined by ICD-11 classification)
* Presence of thoracic or neck pain
* History of previous RF denervation
* Regular use of two or more dependence forming drugs (opioids, gabapentinoids, Benzodiazepines, tricyclics antidepressants and z-drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of either sex, who have been referred for consideration of RF denervation or already found suitable for RF denervation pathway will be eligible for the study. The eligible participant should have nociceptive type, moderate to severe low back pain arising from lumbar facet joints.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
resting state functional connectivity of default mode network | 3 months after treatment
  Any difference between baseline and after successful treatment will be reported as primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom